CLINICAL TRIAL: NCT01352494
Title: A Multi-center Phase II Trial to Evaluate the Efficacy and Safety of Neoadjuvant Chemotherapy With DoceTaxel(Doxotel) and Gemcitabine(Gemcibine)in Locally Advanced Breast Cancer
Brief Title: Neoadjuvant Chemotherapy With Docetaxel and Gemcitabine in Locally Advanced Breast Cancer
Acronym: NeoTG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korean Breast Cancer Study Group (Other)
Responsible Party: Young Jin Suh, Department of Surgery, the Catholic university of Korea, St. Vincent's hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBCSG009
Record Dates: First submitted 2011-05-09; First posted 2011-05-12 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer Stage II; Breast Cancer Stage III
Keywords: locally advanced breast cancer; docetaxel; gemcitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- docetaxel/gemcitabine (Experimental): All the patients are locally advanced breast cancer. Patients with a measurable lesion at chest CT. (at least 1 measurable lesion)
  Interventions: Drug: docetaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: docetaxel — docetaxel - 75 mg/m2, IV (in the vein), every 3 weeks, 4 cycles
  Other Names: Doxotel®
Drug: gemcitabine — gemcitabine - 100 mg/m2, IV (in the vein) on day 1 and 8 day of each 28 day cycle, 4 cycles
  Other Names: Gemcibine®

SUMMARY:
The purpose of this study is to assess the response of docetaxel and gemcitabine in the neoadjuvant setting in women with locally advanced breast cancer.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy is now standard for patients with locally advanced breast cancer, and this method of treatment has been extended to patients with earlier disease without affecting the treatment outcome. This single arm, multicenter phase II study was designed to evaluate the response rate, toxicity, progression free survival and tumor control rate of docetaxel and gemcitabine in the neoadjuvant setting with locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged : 20~70 years
2. World Health Organization (WHO) (Eastern Cooperative Oncology Group [ECOG]) performance status 0-2
3. Patients with measurable lesion assessed by imaging using the RECIST (Response Evaluation Criteria In Solid Tumor) guideline
4. Have given written informed consent and are available for prolonged follow-up

Exclusion Criteria:

1. Patients with previous chemotherapy for recurrent breast cancer
2. Breast cancer recurrence within 12 months after taxane treatment
3. Her-2/neu expression breast cancer
4. Patients with malignancies (other than breast cancer) within the last 5 years, except for adequately treated in situ carcinoma of the cervix or basal cell, squamous cell carcinoma of the skin.
5. Brain metastasis
6. uncontrolled infection, medically uncontrollable heart disease
7. other serious medical illness or prior malignancies
8. Pregnant or lactating women were excluded.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate was assessed by pathologic examination after surgery. | 2 years

SECONDARY OUTCOMES:
Type of surgery (Breast Conserving Rate) | 6 month
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 year
progression free survival | 2 years
quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Young Jin Suh, M.D. Ph.D, Principal Investigator — Department of Surgery, the Catholic university of Korea, St. Vincent's hospital
Locations (1):
- Department of Surgery, the Catholic university of Korea, St. Vincent's hospital, Suwon, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Jeon YW, Kim TH, Youn HJ, Han S, Jung Y, Gwak G, Park YS, Kim JS, Suh YJ. A Multicenter Phase II Trial of Neoadjuvant Chemotherapy with Docetaxel and Gemcitabine in Locally Advanced Breast Cancer. J Breast Cancer. 2017 Dec;20(4):340-346. doi: 10.4048/jbc.2017.20.4.340. Epub 2017 Dec 19. PMID 29285038